CLINICAL TRIAL: NCT00872638
Title: The Effect of Wound Edge Eversion on Cosmesis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of participation
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Adam Singer, research director, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 20076828
Record Dates: First submitted 2009-03-28; First posted 2009-03-31 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Surgical Incisions
Keywords: wound edge eversion; cosmetic outcomes; surgical incisions
MeSH Terms: conditions — Surgical Wound | interventions — Automated Facial Recognition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Procedure: Eversion
- 2 (Active Comparator)
  Interventions: Procedure: Approximation

INTERVENTIONS:
Procedure: Eversion — Surgical incisions will be closed in such a manner so as to evert the wound edges.
  Other Names: mattress sutures
  Arms: 1
Procedure: Approximation — Surgical incisions will be closed in such a manner so that wound edges are approximated exactly, i.e. without eversion.
  Other Names: simple suture
  Arms: 2

SUMMARY:
Aesthetic appearance of repaired incisions is very important to surgical patients. It has been stated that if the edges of a wound are closed in such a manner that will result in eversion, or pouting of the edges that the end cosmetic result will be superior when compared to wound edges that are simply approximated. The purpose of this study is to compare cosmetic outcomes of incisions that are closed with everted edges to those in which the edges are simply approximated.

DETAILED DESCRIPTION:
Surgical incisions will be split into two halfs and each half will be randomized to standard or everting sutures. 3 months later the cosmetic outcome of the healed wounds will be determined using a validated scar evaluation scale.

ELIGIBILITY:
Inclusion Criteria:

* age over 18.
* able to consent.
* scheduled for elective plastic or cardiothoracic surgery.

Exclusion Criteria:

* history of keloids, hypertrophic scarring, diabetes, or peripheral vascular disease.
* those requiring systemic steroids or undergoing chemotherapy, and those unable or unwilling to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Cosmetic result of surgical incision as measured by VAS scale | 1 year

SECONDARY OUTCOMES:
Cosmetic Results as measured by the Stony Brook Scar Scale | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Adam Singer, MD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University Medical Center, Stony Brook, New York, United States